CLINICAL TRIAL: NCT05053750
Title: TAME: A Pilot Study of Weekly Paclitaxel, Bevacizumab, and Tumor Associated Macrophage Targeted Therapy (Zoledronic Acid) in Women With Recurrent, Platinum-resistant, Epithelial Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gateway for Cancer Research (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0694; NCI-2021-10703 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-09-15; First posted 2021-09-22 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Epithelial Ovarian; Fallopian Tube; Primary Peritoneal Cancer
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paclitaxel (Experimental)
  Interventions: Drug: Paclitaxel/Bev (control)
- Bevacizumab (Experimental)
  Interventions: Drug: Paclitaxel/Bev + ZA (experimental)

INTERVENTIONS:
Drug: Paclitaxel/Bev (control) — Given by PO
  Other Names: Taxol
  Arms: Paclitaxel
Drug: Paclitaxel/Bev + ZA (experimental) — Given by PO
  Arms: Bevacizumab

SUMMARY:
This is a randomized pilot trial of weekly paclitaxel and bevacizumab with or without zoledronic acid in women with platinum-resistant epithelial ovarian cancer with 1-2 prior regimens for recurrence.

DETAILED DESCRIPTION:
Primary Objective:

-To assess macrophage counts by image cytometry in women with platinum resistant ovarian cancer treated with weekly paclitaxel/bevacizumab and ZA relative to weekly paclitaxel/bevacizumab. The primary endpoint is the percentage changes in macrophage count from baseline to after 2 cycles of therapy.

Secondary Objective:

* To estimate the progression free survival (PFS) of combination weekly paclitaxel/bevacizumab and ZA relative to weekly paclitaxel/bevacizumab in women with platinum-resistant recurrent ovarian cancer
* To evaluate toxicity of the two arms
* To assess objective response and duration of response by RECIST 1.1
* To estimate overall survival

Exploratory Objective

To assess differential effects from baseline, within and between patient treatment cohorts, on macrophage and hypoxia markers, CSF1/R and MHCII, plasma biomarker (VEGF, VEGFR, IL6, IL8, FGF, PDGFAA), tumor and macrophage-derived exosomes, and single-cell level changes.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all the following criteria apply within 28 days of starting study treatment. be assessed

1. Ability to provide signed informed consent
2. Age ≥ 18 years at time of study entry
3. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
4. Histologically confirmed and documented platinum refractory* or platinum resistant** high grade epithelial ovarian cancer to include: adenocarcinoma NOS, clear cell adenocarcinoma, endometrioid adenocarcinoma, malignant Brenner's tumor, mixed epithelial carcinoma, serous adenocarcinoma, transitional cell carcinoma, and undifferentiated carcinoma. * Platinum refractory is defined as progression during platinum-containing therapy or within 4 weeks of last dose. ** Platinum resistant is defined as relapse-free interval 1-6 months of a platinum-containing therapy
5. Prior Therapy: Unlimited prior systemic therapies are allowed.
6. ECOG performance status of 0-1
7. Life expectancy > 12 weeks
8. Adequate normal organ and marrow function as defined below.

   1. Hemoglobin ≥9.0 g/dL.
   2. Absolute neutrophil count (ANC) > 1500/mm3

      .
   3. Platelet count ≥100 x 109

      /L
   4. Serum bilirubin ≤1.5 x ULN. This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
   5. AST (SGOT)/ALT (SGPT) ≤2.5 x ULN unless liver metastases are present, in which case it must be ≤5x ULN.
   6. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

   Creatinine CL (mL/min)

   = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
9. Evidence of post-menopausal status or negative serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   1. Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the postmenopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   2. Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply within 28 days of starting study treatment.

1. Nonepithelial tumors including carcinosarcomas. Mucinous ovarian cancers. Ovarian tumors with low malignant potential or low-grade epithelial tumors.
2. Patients who have received anti-VEGF targeted therapy (alone or in combination with chemotherapy or other biological agents) for recurrent disease and have progressed on that therapy or within 6 months of discontinuation of that therapy. Prior bevacizumab in the upfront setting is permitted.
3. History of other clinically active malignancy within 5 years of enrollment, except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix or breast, or early stage endometrial cancer (stage IA/B, Grade 1 or 2, endometrioid histology).
4. Patients with known or suspected conditions likely to increase gastrointestinal toxicity, such as, inflammatory bowel disease, bowel obstruction, history of bowel obstruction or overt bowel involvement by tumor.
5. History of bowel obstruction, including sub-occlusive disease, related to the underlying disease and history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess. Evidence of recto-sigmoid involvement by pelvic examination or bowel involvement on CT scan or clinical symptoms of bowel obstruction.
6. Patients who are pregnant or lactating.
7. Radiation, chemotherapy, or immunotherapy or any other anticancer therapy ≤2 weeks prior to cycle 1 day 1.
8. Major surgery (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within four weeks before Day 1.
9. Unstable cardiovascular function:

   * ECG abnormalities requiring treatment, or
   * congestive heart failure (CHF) of NYHA Class ≥3, or
   * myocardial infarction (MI) within 3 months.
10. Uncontrolled infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose; patients with controlled infection or on prophylactic antibiotics are permitted in the study.
11. Known active hepatitis A, B, or C infection; or known to be positive for HCV RNA or HBsAg (HBV surface antigen); Known to be HIV seropositive
12. Any underlying condition that would significantly interfere with the absorption of an oral medication.
13. Grade >2 peripheral neuropathy at baseline (within 14 days prior to cycle 1 day 1).
14. Patients with urine dipstick for proteinuria >2+. Patients with ≥2+ proteinuria on baseline dipstick analysis should undergo a 24-hour urine collection and must demonstrate ≤1 g of protein in the 24-hour urine. Alternatively, proteinuria testing can be performed according to local standards.
15. Serious psychiatric or medical conditions that could interfere with treatment;
16. Participation in an investigational anti-cancer study within 3 weeks prior to Cycle 1 Day 1
17. Concurrent therapy with approved or investigational anticancer therapeutic other than steroids.
18. Patients with coagulation problems and active bleeding within 4 weeks prior to C1D1 (peptic ulcer, epistaxis, spontaneous bleeding)
19. Patients with symptomatic brain lesions
20. For women who are not postmenopausal (<12 months of non therapy-induced amenorrhea, with no identified cause other than menopause) and have not undergone surgical sterilization (removal of ovaries and/or uterus): agreement to remain abstinent (refrain from heterosexual intercourse) or use two adequate non hormonal methods of contraception, including at least one method with a failure rate of <1% per year, during the treatment period and for at least 4 months after the last dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
To assess macrophage counts by image cytometry in women with platinum resistant ovarian cancer treated with weekly paclitaxel/bevacizumab and ZA relative to weekly paclitaxel/bevacizumab | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Westin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT05053750/ICF_000.pdf